CLINICAL TRIAL: NCT06270745
Title: ICG Anastomotic Control in Digestive System Surgery
Status: Recruiting | Type: Observational
Sponsor: Shandong Linglong Yingcheng Hospital (Network)
Responsible Party: Sponsor
Other Study IDs: sdycllyy001
Record Dates: First submitted 2024-02-14; First posted 2024-02-21 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Surgical Anastomosis
Keywords: Surgical Anastomosis,Anastomotic leak ,perfusion
MeSH Terms: interventions — Indocyanine Green

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Indocyanine Green: Indocyanine green infusion during digestive system surgery
  Interventions: Drug: indocyanine green
- non-Indocyanine Green: No indocyanine green infusion during digestive system surgery
  Interventions: Drug: indocyanine green

INTERVENTIONS:
Drug: indocyanine green — Whether to use ICG to assess anastomotic perfusion during digestive system surgery

SUMMARY:
This was a parallel single-center retrospective cohort study conducted at Linglong Yingcheng Hospital, Shandong, China. The purpose of this study was to investigate the effect of indocyanine green (ICG) on patients undergoing digestive system surgery (subtotal gastrectomy, partial hepatectomy, transverse colectomy, left colectomy, including sigmoid resection, and splenic colic resection). ) of anastomotic leakage (AL). Secondary objectives were to detect and study the impact of various risk factors on AL and on morbidity and surgical performance within 30 days of surgery.

DETAILED DESCRIPTION:
This was a parallel single-center retrospective cohort study observing a series of consecutive patients who underwent colorectal surgery at our institution between January 1, 2018, and December 31, 2023.

The primary endpoint of the study is AL at 30 days, and the secondary endpoint is postoperative morbidity of Clavien-Dindo score ≥ III within 30 days after surgery, including readmission and redo surgery, lymph node disease in patients with neoplastic disease Harvest, surgical site infection, laparoscopic surgery rate, and protected stoma rate.

According to the American Joint Committee on Cancer (AJJC) 8th edition, gender, body mass index, smoking, diabetes, cardiovascular disease, and tumor stage will be considered confounding factors in the development of AL.

A patient electronic database will be collected from medical records extracted from surgical logs and each digital medical record will be scanned to include perioperative outcomes and post-operative follow-up for 30 days after surgery, final readmission to the emergency room or any other department based on The following inclusion criteria, performed in the specialist ward of our local health institution: elective surgery, left colon segmental surgery: splenic colic resection, transverse colic resection and left hemicolectomy, defined as left hemicolectomy, low Mesenteric artery ligation and sigmoid resection, regardless of benign or malignant pathology, minimum 30 days of postoperative follow-up (available from medical documentation), primary colostomy or colorectal anastomosis with or without prophylactic ostomy ) and age of adulthood.

Exclusion criteria were distal colostomy without anastomosis after removal step, extended transverse right hemicolectomy, left hemicolectomy with high vascular ligation, resection of associated bowel or other viscera (ie, tumor infiltration), previous colic Surgery, synchronous tumors, failure to report vessel ligation in surgery form details, lack of medical record reporting of primary outcome, stage IV cancer, American Society Of Anestheasiologists (ASA) IV, under 18 years of age, and emergencies.

Reconstruction times vary with different anastomoses (colostomy or colorectal), techniques (staplers or hand suturing), and connections (side to side, side to end, end to side, or end to end).

Since 2018, our institute has been using ICG fluorescence laparoscopy, using a near-infrared (NIR) light source and a special oscilloscope and camera equipped with a xenon lamp; ICG is available as a sterile water-soluble lyophilized powder (Diagnostic Green® GmbH) . ICGICG fluorescence laparoscopy is routinely used in daily practice, following the following protocol: after specimen resection and before anastomosis, both colonic stumps or the colon and rectal stumps are examined with 5 cc of ICG 25 mg diluted in 10 cc of sterile aqueous solution .

Statistical analysis and sample size:

Quantitative variables will be described by mean ± standard deviation or median and IQR, and qualitative variables will be described by absolute frequency and percentage frequency. All continuous variables will be checked for normality. Comparisons of covariates will be performed using the Pearson X2 test or Fisher's exact test (for categorical variables) and the t test or Mann Whitney test (for continuous variables). Univariate analysis will be performed using logistic regression to examine the association of each predictor variable with anastomotic leak events. Next, variables with p<0.1 were considered for inclusion in the multivariable regression model. For each risk factor, the odds ratio is shown along with the associated confidence interval. All analyzes will be performed using spss version 27.0 statistical software with two-sided significance tests and a 5% significance level.

ELIGIBILITY:
Inclusion Criteria:

* elective setting of surgery
* digestive system surgery for benign or malignant pathology
* 30 days of post-operative follow-up at least available from medical documentation
* primary colo-colic or colo-rectal anastomosis with or without preventing ostomy
* more than 18 years old, less than 90 years old

Exclusion Criteria:

* terminal colonic stoma without anastomosis creation after demolitive step
* extended transverse right hemicolectomy
* left hemicolectomy with high vascular ligation
* associated bowel or another splanchnic resection (i.e. neoplastic infiltration)
* previous colic surgery
* synchronous neoplasm
* not reporting in operating form details about vascular ligation
* lack in reporting in medical records of primary outcomes
* stage IV cancer
* ASA IV
* less than 18 years old, more then 90 years old
* emergency setting

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A consecutive series of patients underwent digestive system surgery at our institution between January 1, 2018, and July 31, 2023
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Anastomotic leak at 30 days | 30 days
  Anastomotic leak (a defect of intestinal wall at anastomotic site leading to a communication between the intra- and extraluminal compartments)at 30 days: abdominal CT scan IV and a Clavien Dindo Score ≥III

SECONDARY OUTCOMES:
Post-operative morbidity | 30 days
  Clavien-Dindo score ≥III within 30 days from surgery including readmission and redo-surgery, harvested nodes for patients with neoplastic disease, Surgical Site Infection, rate of laparoscopic surgical procedure and rate of protection stoma.

CONTACTS AND LOCATIONS:
Overall Officials: Xuan Qiu, MD, Principal Investigator — Shandong Linglong Yingcheng Hospital
Locations (1):
- Shandong Linglong Yingcheng Hospital, Yantai, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Qiu X, Kashchenko VA, Zavrazhnov AA, Lankov TS, Ye L, Strizheletsky VV, Smirnov GA. Deep impact analysis of surgical strategy changes guided by indocyanine green fluorescence angiography in laparoscopic low anterior resection for rectal cancer. Int J Colorectal Dis. 2026 Jan 3;41(1):7. doi: 10.1007/s00384-025-05065-8. PMID 41483178